CLINICAL TRIAL: NCT05837754
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Assess the Gut Health Effects of Oil Compound on Healthy Adults
Brief Title: A Study to Assess the Gut Health Effects of Oil Compound on Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: JR/220801/OC/GH
Record Dates: First submitted 2023-03-23; First posted 2023-05-01 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Gut Health

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled, parallel group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Stratified block randomization, Sequentially numbered, sealed, opaque envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C8-C12 (Active Comparator): 5-15mL (one teaspoon to one tablespoon) once or twice a day. The participants will be dispensed a 5 ml pipette for consuming the IP
  Interventions: Other: C8-C12
- Placebo (Placebo Comparator): 5-15mL (one teaspoon to one tablespoon) once or twice a day. The participants will be dispensed a 5 ml pipette for consuming the IP
  Interventions: Other: Placebo

INTERVENTIONS:
Other: C8-C12 — 5-15mL (one teaspoon to one tablespoon) once or twice a day. The participants will be dispensed a 5 ml pipette for consuming the IP.
  Arms: C8-C12
Other: Placebo — 5-15mL (one teaspoon to one tablespoon) once or twice a day. The participants will be dispensed a 5 ml pipette for consuming the IP.
  Arms: Placebo

SUMMARY:
The present study is a randomized, placebo-controlled, double-blind, parallel group study to assess the gut health effects of IP as compared to a placebo in normal, overweight and obese individuals experiencing gut issues. Approximately 94 will be randomized into 1:1 ratio to either receive IP or Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with the age ≥18 and ≤60 years with active lifestyle, moderate physical activity level as per International Physical Activity Questionnaire - Short Form (IPAQ-SF)
* BMI of ≥ 18 - ≤ 34.9 kg/m2
* Having at least three of the following five metabolic risk factors:

  1. Waist circumference > 102 cm (40 inches) for men and > 88 cm (35 inches) for women;
  2. Fasting triglycerides >150 mg/dL
  3. Blood pressure ≥130 mm Hg (Systolic Blood Pressure) and/or ≥85 mm Hg (Diastolic Blood Pressure);
  4. Fasting blood glucose ≥ 100 mg/ dl
  5. Fasting HDL cholesterol level less than 40 mg/dl (men) or 50 mg/dl (women)
* SGOT, SGPT ≤ 2 times the upper normal limit.
* Creatinine levels ≤ 1.5 times the upper normal limit.
* Willing to complete all study procedures including study related questionnaires and comply with study requirements.
* Willing to abstain from other supplements or medication.
* Ready to give voluntary, written, informed consent to participate in the study.
* Evidence of abnormal stool consistency (at least one day every week indicating constipation or diarrhoea) as determined by Bristol Stool Scale in the last 3 months.
* No self-reported physical/mental disabilities or gastrointestinal conditions.
* No antibiotic usage within the last 30 days.
* History of stable weight over the last 6 months (<10% change).
* Willing to maintain current dietary and exercise habits, aside from any changes to be made per the study exercise protocol.

Exclusion Criteria:

* Pure vegetarians who do not consume chicken, fish and/or egg.
* Smokers
* Presence of unstable, acutely symptomatic, or life-limiting illness.
* Subjects with uncontrolled hypertension with systolic blood pressure ≥160 and diastolic blood pressure ≥100 mm Hg.
* Subjects with uncontrolled Type II Diabetes Mellitus with FBG ≥ 126 mg/ dl
* Neurological conditions causing functional or cognitive impairments.
* Unwillingness or inability to be randomized to one of two intervention groups.
* Bilateral hip replacements.
* History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders that, in the judgment of the Investigator, would interfere with the participant's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the participant at undue risk.
* History or presence of Irritable Bowel Syndrome as per Rome IV criteria. [Diagnostic criteria* Recurrent abdominal pain on average at least 1 day/week in the last 3 months, associated with two or more of the following criteria:

  1. Related to defecation.
  2. Associated with a change in frequency of stool.
  3. Associated with a change in form (appearance) of stool. *Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis]
* Use of any psychotropic medication within four weeks of screening and throughout the study.
* Use of antibiotics or signs of active systemic infection at the time of screening. Treatment visits will be rescheduled to the subject to wash off the antibiotic for at least five days prior to any test visit.
* Subject states they regularly consume supplemental enzymes and are unwilling to stop at least one week prior to screening and throughout the study. Supplemental enzymes may include standalone enzyme supplements, probiotic supplements with enzymes, and any medications containing enzymes.
* Subject states they regularly consume probiotic, prebiotic, energy and mood enhancing supplements supplements and are unwilling to stop at least one week prior to screening and throughout the study. Supplemental probiotics may include standalone probiotic supplements, vitamins with probiotics, and any foods supplemented with probiotics
* Subject states they are currently being prescribed (by primary care physician or other health professional) medication or using an over-the-counter product that in the opinion of the study physician will have an effect on food digestion or nutrient absorption during the study.
* Exposure to any non-registered drug product within 3 months prior to the screening visit.
* Unable/unwillingness to complete study specific diaries (digital/paper-based).
* Current use of the following medications: monoamine oxidase inhibitors, prescription or herbal weight loss medications/ dietary supplement.
* Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
* Heavy alcohol drinkers defined as follows:

For men, consuming more than 4 drinks on any day or more than 14 drinks/week For women, consuming more than 3 drinks on any day or more than 7 drinks/week

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of the Investigational Product (IP) on | Day 56
  Gut permeability by assessing the levels of Lipopolysaccharide Binding Protein at day 56 from baseline.

SECONDARY OUTCOMES:
To assess the effect of the of IP on Daily energy levels using Visual Analogue Scale - Fatigue | Day 0,1,2,3,4,5,28 and 56
  The respondents will be asked to denote the severity of their fatigue at the present moment by placing a mark on a line extending from "no fatigue" to "fatigue as bad as could be." Higher scores on the scale are indicative of more severe fatigue.
To assess the effect of the of IP on Fatigue Severity Scale (FSS) | Day 0, 28 and 56
  The FSS is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Grading of each item ranges from 1 to 7, where 1 indicates strong disagreement and 7 indicates strong agreement, and the final score represents the mean value of the 9 items.
To assess the effect of the of IP on Immunomodulation using IFN-γ. | Day 0, 28 and 56
  The serum levels of the IFNγ in healthy lean population was 10.83 ± 5.81 pg/ml and in obese population was 9.35 ± 5.14 pg/ml.
To assess the effect of the of IP on Inflammation using TNF-α, IL-6 and IL-10 | Day 0, 28 and 56
  The recommended reference ranges of serum TNF-α is upto 10 pg/mL. The reported values for serum IL-6 in the blood of healthy individuals varied between 0 and 15 pg/ml. The detection ranges of IL-10 is 7.8 pg/ml to 500 pg/ml. The reported values for serum IL-10 in the blood of healthy controls upto 5 pg/ml.
To assess the effect of the of IP on Stress as assessed by the change in the Perceived Stress Scale. | Day 0, 28 and 56
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
To assess the effect of the of IP on Quality of life using Digestive Associated Quality of Life Questionnaire (DQLQ). | Day 0, 28 and 56
  The DQLQ includes 9 statements. The total score represents the sum of the responses to the 9 statements with possible scores ranging from 0 to 9. A higher score indicates a lower (worse) digestion-associated QOL.
To assess the effect of the of IP on Satiety as assessed by the change in the Three-Factor Eating Questionnaire-R18 (TFEQ-R18). | Day 0, 28 and 56
  It is an 18 item questionnaire, where the responses are scored on a four-point scale (1 = definitely false, 2 = mostly false, 3 = mostly true, 4 = definitely true) and summed, except the question no. 18 where the scoring will be done on an eight-pointer scale. The higher score depicts the high degree of occurrence of the behavior, and higher levels of eating disturbances.
To assess the effect of the of IP on Mood states using Mood and Feelings Questionnaire (MFQ) | Day 0, 28 and 56
  Responses are rated on a 3-point scale. Total scores range from 0 to 26, with a score ≥12 commonly used in the literature to indicate clinically significant depression.
To assess the effect of the of IP on Clinical Responders as assessed by the number of participants achieving normal stool consistency using Bristol stool form scale (BSFS). | Day 0 and 56
  A tool that categorises the stool into one of seven stool types ranging from type 1 (hard lumps) to type 7 (watery diarrhoea).
To assess the effect of the of IP on Gut microbiome diversity using | Day 0 and 56
  16s RNA sequencing

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - Apex Hospital, Ahmedabad, Gujarat
  - Aman Hospital and Research Centre, Vadodara, Gujarat
  - Hira Mongi Navneet Hospital, Mulund East, Maharashtra
  - Shantaee Nursing Home, Mumbai, Maharashtra
  - Sangvi Multispeciality Hospital, Pune, Maharashtra
  - Lifepoint Multispeciality Hospital, Pune, Maharashtra
  - Maharaja Agrasen Superspeciality Hospital, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: No